CLINICAL TRIAL: NCT06993753
Title: Queensland Infant Birth Dose RSV Immunisation Program 2024 - Duration of Protection and Impact
Brief Title: Duration of Protection of Nirsevimab Against Hospitalisation for Respiratory Syncytial Virus Infection
Status: Active, not recruiting | Type: Observational
Sponsor: Griffith University (Other)
Responsible Party: Principal Investigator, Asmaa El-Heneidy, Dr, Griffith University
Other Study IDs: 2024/851; VAS00012 (Other Grant/Funding Number: Sanofi Pasteur S.A)
Record Dates: First submitted 2025-05-19; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-02

CONDITIONS: Respiratory Syncytial Viral (RSV) Infections
Keywords: Respiratory syncytial virus; Case control; monoclonal antibody; nirsevimab
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- RSV hospitalised infant: Description: Cases (RSV hospitalised infant) will be children born in Queensland from 15 April 2024 to 14 April 2025 who are hospitalised with a RSV-related condition prior to 14 April 2026. Nirsevimab receipt will be extracted from hospital's electronic medical records and linked to hospitalisation data by the Queensland Health Data Linkage Unit.
- Non-RSV hospitalised infant: Description: Controls (Non-RSV hospitalised infant) will be drawn from the set of infants who are admitted to the same hospital in a 5:1 ratio, and matched on age and sex using the Queensland Perinatal Data Collection. Nirsevimab receipt will be extracted from hospital's electronic medical records and linked to hospitalization data by the Queensland Health Data Linkage Unit.

SUMMARY:
Respiratory syncytial virus (RSV) is a leading cause of hospitalizations for acute lower respiratory tract infection (LRTI) in infants. In Australia approximately 1.5% of infants are hospitalized due to RSV, 80% of whom are born full-term and are otherwise healthy. Two randomized trials have used a seasonal implementation strategy to show nirsevimab, a long-acting monoclonal antibody, has sustained efficacy against RSV LRTI hospitalizations in the first 150-180 days after administration. Nirsevimab has been approved in many countries for the prevention of RSV-LRTI in neonates and infants. However, the protection offered by nirsevimab beyond 180 days remains unknown. Queensland is a large Australian state spanning the tropical and sub-tropical climate zones, where RSV circulates year-round. The Queensland government publicly funded nirsevimab for all infants at birth from 15 April 2024. The aim of this study is to estimate the duration of effectiveness of nirsevimab against RSV-related hospitalizations.

A case-control study will be conducted using routinely collected linked data. Cases will be children born in Queensland from 15 April 2024 to 14 April 2025 who are hospitalised with an RSV-related condition prior to 14 April 2026. Controls will be drawn from the set of infants who are admitted to the same hospital in a 5:1 ratio, and matched on age and sex using the Queensland Perinatal Data Collection. Nirsevimab receipt will be extracted from hospital's electronic medical records and linked to hospitalization data by the Queensland Health Data Linkage Unit. Duration of protection against RSV-related hospitalisation due to nirsevimab will be assessed using multivariable logistic regression model accounting for matching and adjusting for confounding variables.

This case-control study will determine the level and duration of protection offered by nirsevimab in a region with year-round RSV circulation and inform future prevention strategies. Interim analysis is expected to be available at the time of the conference, allowing for early dissemination of this first evidence about nirsevimab duration of protection beyond 180 days.

Funding: From Sanofi and AstraZeneca through a collaboration grant.

ELIGIBILITY:
Inclusion Criteria: Any infant born between 15 April 2024 and 30 April 2025 and hospitalized for any reason between 15 April 2024 and 30 April 2026.

Exclusion Criteria: Infants who admitted to hospitals with an elective admission. ((i.e. admissions that are planned ahead of time, such as scheduled surgeries or other pre-arranged medical procedures).

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Our study population will consist of all infants born in Queensland between 15 April 2024 and 30 April 2025 and hospitaliszed for any reason between 15 April 2024 and 30 April 2026.
  Cases will be All infants born in Queensland between 15 April 2024 and 30 April 2025 who were admitted to any hospital in Queensland (public and private) between 15 April 2024 and 30 April 2026 with a respiratory related principle or other diagnosis (ICD codes J21.0, J20.5, J12.1, B97.4). Controls will be defined as infants admitted to the same hospital that do not have a diagnosis of (ICD codes J21.0, J20.5, J12.1, B97.4) and that the admission is not an elective admission.
  For each included case, five controls (where possible) matched on month of birth and sex will be requested to enable appropriate comparison.
Sampling Method: Non-Probability Sample
Enrollment: 4350 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
The duration of effectiveness of nirsevimab against RSV-related hospitalizations. | From mid April 2024 to mid April 2026

SECONDARY OUTCOMES:
Estimate the quantities of the laboratory confirmed RSV hospitalization length of stay and paediatric intensive care unit admission that were prevented by a 12-month year-round nirsevimab immunization program in Queensland infants. | From mid April 2024 to mid April 2026
Estimate the quantities of all cause acute respiratory hospitalization and PICU admissions that were prevented by nirsevimab immunization program in Queensland infants | From mid April 2024 to mid April 2026
Estimate the quantities of all death from RSV-related illness that were prevented by a 12-month year-round nirsevimab immunization program in Queensland infants | From mid April 2024 to mid April 2026
Evaluate the impact of nirsevimab on the cost of hospital services in Queensland, Australia | From mid April 2024 to mid April 2026

CONTACTS AND LOCATIONS:
Locations (1):
- Griffith University, Gold Coast, Queensland, Australia

IPD SHARING:
Plan to Share IPD: Undecided